CLINICAL TRIAL: NCT06469879
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of TQB2450 Combined With Anlotinib as Maintenance Therapy in Patients With Limited-stage Small Cell Lung Cancer
Brief Title: A Clinical Study of TQB2450 Combined With Anlotinib in Limited-Stage Small Cell Lung Cancer Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB2450-ALTN-III-01
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Small Cell Lung Cancer Limited Stage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450+Anlotinib (Experimental): TQB2450 injection: 1200 mg/time, intravenous infusion, day 1, every 3 weeks (Q3W); Anlotinib hydrochloride capsules: 8 mg/time, once a day (QD), for 2 weeks, stop for 1 week, oral before breakfast; (The starting dose of anlotinib hydrochloride is 8 mg, and an upward adjustment to 10 mg is allowed after two cycles.)
  Interventions: Drug: TQB2450+Anlotinib
- TQB2450 placebo + anlotinib placebo (Placebo Comparator): TQB2450 injection placebo: 0 mg/time, intravenous drip, day 1; anlotinib hydrochloride capsule placebo: 0 mg/time, once a day (QD), for 2 consecutive weeks, stop for 1 week, oral administration before breakfast.
  Interventions: Drug: TQB2450 placebo + Anlotinib placebo

INTERVENTIONS:
Drug: TQB2450+Anlotinib — TQB2450 injection test group, 1200 mg/time, strength: 600mg/20 mL, intravenous drip, day 1, every 3 weeks. Anlotinib hydrochloride capsules: 8 mg/time, strength: 10mg/capsule, 8mg/capsule, 6mg/capsule., 1 time a day (QD), continuous use for 2 weeks and stop for 1 week.
  TQB2450 Injection Placebo (control group): 0 mg/time, strength: 0mg/20 mL, Intravenous Drip, Day 1, every 3 weeks. Anlotinib hydrochloride capsule placebo: 0 mg/time, strength: 0mg/capsule, 1 time a day (QD), continuous use for 2 weeks and stop for 1 week.
  Arms: TQB2450+Anlotinib
Drug: TQB2450 placebo + Anlotinib placebo — No drug substance is contained
  Arms: TQB2450 placebo + anlotinib placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled phase III clinical study to evaluate the efficacy and safety of TQB2450 in combination with anlotinib as maintenance therapy in patients with limited-stage small cell lung cancer who have not progressed after chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent, and the compliance was good;
* Age: 18~75 years old (when signing the informed consent form); Eastern Cooperative Oncology Group Performance Status score: 0-1 points; expected survival of more than 6 months; weight > 40 kg;
* Pathologically confirmed patients with limited stage small cell lung cancer (according to the Veterans Administration Lung Study Group (VALG) stage);
* There was no evidence of metastatic disease by diagnostic quality enhanced CT of the neck, chest, abdomen, and pelvic cavity, and craniocerebral plain scan plus enhanced MRI (PET-CT is recommended before chemoradiotherapy. Bone scan should be performed if PET-CT is not performed before chemoradiotherapy. PET-CT must be performed during the screening period after chemoradiotherapy to rule out metastasis.);
* It is anticipated that no tumor resection will be required during the study（Patients who are not suitable for surgery or those who do not want surgery can be treated);
* Receive the chemoradiotherapy regimen prescribed below, unless an alternative is acceptable after consultation with the investigator:

  1. Four cycles of platinum-containing chemotherapy with concurrent or sequential radiotherapy were received, and these treatments had to be completed within 1 to 42 days of randomization and the first administration of the study drug;
  2. According to the standard treatment regimen at each study center, chemotherapy regimens must contain cisplatin/carboplatin drugs and etoposide administered intravenously
  3. For the standard Quaque Die radiotherapy regimen, the total radiation dose received was 60 Gy±10% (6-week regimen), and for the hyperfractionated Bis in die radiotherapy regimen, the total radiation dose received was 45 Gy (3-week regimen), and the dose was calculated based on the planned target area (PTV). Research centers are encouraged to follow the following doses of radiation to organs at risk：

  c.1 Average lung dose <20 Gy and/or V20 must be <35% c.2 Cardiac V50 <25% d. If synchronous Cardiac resynchronization therapy is used, chest radiotherapy must be started no later than the first day of the 3rd cycle of chemotherapy; e. If sequential radiotherapy is used, thoracic radiotherapy should be preceded by at least 2 cycles of induction chemotherapy, with no more than 35 days between the end of the chemotherapy cycle and the start of radiotherapy;
* Precision radiotherapy techniques such as three-dimensional conformal radiotherapy, conformal intensity modulated radiotherapy and tomographic radiotherapy are adopted;
* Patients receiving radical platinum-based chemoradiotherapy must achieve complete response, partial response, or stable disease without disease progression;
* Prophylactic brain radiotherapy (PCI) is permitted according to the judgment of the investigator and the standard treatment at each study center, and must be performed after the completion of Cardiac resynchronization therapy, but it is allowed to be targeted at the last chemotherapy;
* The patient provided tumor tissue as far as possible for Programmed cell Death ligand 1 (PD-L1) expression level determination. Any available tumor tissue sample can be submitted: histology or cytology (if tissue samples are not available). Pathology reports of these specimens must also be provided;
* The patient was confirmed to have at least one measurable lesion according to RECIST 1.1 criteria prior to chemoradiotherapy;
* Having an adequate Pulmonary function test, defined as Forced expiratory volume in one second > 50% of predicted normal expiratory volume and Diffusing capacity of the lung for carbon monoxide (DLCO) > 40% of predicted normal. For subjects without diffusing capacity of the lungs for carbon monoxide measurements, adequate oxygen transport is considered if the pulse oxygen saturation (O2 saturation) measured in indoor air is ≥ 90%.

Exclusion Criteria:

* Tumor disease and history

  1. Present or present with other malignant tumors within 3 years. The following two conditions can be included: 5 consecutive years of disease-free survival (DFS) without any treatment for other malignancies; Cured of thyroid cancer, Cervical carcinoma in situ, Non-melanoma skin cancer and superficial bladder tumors【Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basal membrane)】;
  2. Complex small cell lung cancer confirmed by histopathology or cytopathology;
  3. Subjects with known central nervous system metastatic and/or cancerous meningitis;
  4. Malignant pleural effusion and pericardial effusion；
  5. Patients whose imaging (CT or MRI) shows that the tumor has invaded an important blood vessel or who are judged by the investigator to be highly likely to invade an important blood vessel during subsequent studies and cause a fatal hemorrhage;
* Previous antitumor therapy

  1. Within 2 weeks prior to the start of the study treatment, the patients were treated with proprietary Chinese medicines with anti-tumor indications specified in theNational Medical Products Administration approved drug specification (Including compound cantharidin capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Brucea oil injection/capsule, Xiaoaiping tablet/injection, Huachansu capsule and so on);
  2. Patients who have received immunomodulatory drugs (e.g., interleukin-2, thymosin, lentinan, etc.) within 30 days before starting treatment；
  3. Prior treatment with an anti-programmed death-1, anti-Programmed cell death 1 ligand 1, or anti-Programmed death ligand-2 drug or against another irritating or co-inhibitory T cell receptor (e.g. cytotoxic T lymphocyte-associated antigen-4, OX 40, TNFRSF9, 4-1BB)；
  4. In the past, he used bevacizumab,Anlotinib, Apatinib and other anti-angiogenic drugs；
  5. Received more than 4 courses of chemotherapy。Chemotherapy regiments other than etoposide and platinum are not allowed；
  6. Unmitigated toxic effects above Common Terminology Criteria for Adverse Events grade 1 due to any prior treatment（Hearing loss, hair loss, fatigue and abnormal lymphocyte count due to prior chemoradiotherapy were not included）；
  7. Subjects with ≥ grade 2 pulmonary inflammation after prior chemoradiotherapy;
* Combined disease and history

  1. Cirrhosis, active hepatitis*:

     Active hepatitis（Hepatitis B reference: HBsAg positive, and Hepatitis B virus DNA detection value exceeds the upper limit of normal value; Hepatitis C reference: Hepatitis C virus antibody positive and Hepatitis C (HCV) virus titer test values above the upper limit of normal); Note: Participants who are eligible for enrollment, hepatitis B surface antigen positive or core antibody positive, and hepatitis C patients need continuous antiviral therapy to prevent virus activation.
  2. Patients with renal failure requiring hemodialysis or peritoneal dialysis have pre-existing or existing nephrotic syndrome or chronic nephritis
  3. Cardio-cerebrovascular abnormalities:

  c.1 Have grade 2 myocardial ischemia or myocardial infarction, arrhythmia (including QT Interval Correction ≥450ms in men, QT Interval Correction ≥470ms in women), and grade 2 congestive heart failure (NYHA rating); c.2 Severe arterial/venous thrombosis events, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc., occurred within 6 months; c.3 After two or more medications, blood pressure control remained unsatisfactory (systolic ≥150 mmHg or diastolic ≥90 mmHg) d. History of immunodeficiency: d.1 A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; d.2 Active autoimmune disease requiring systemic treatment (such as use of disease-modifying drugs, corticosteroids, or immunosuppressants) occurred within 2 years prior to study treatment initiation(Such as, but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; Subjects with asthma requiring medical intervention with bronchodilators were not included). Hormone replacement therapy (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) may not be considered systemic treatment; e. Have been diagnosed with an immune deficiency or are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose >10mg/ day prednisone or other therapeutic hormone) and continue to use within 2 weeks prior to initial administration; f. Patients with active tuberculosis within 1 year prior to enrollment; Participants with a history of active pulmonary tuberculosis infection before 1 year were required to provide clear evidence of cure. If tuberculosis was suspected during the screening period, the patients could be enrolled only after being excluded by chest radiography or chest CT, sputum and clinical symptoms;
* Study live attenuated vaccine vaccination history within 28 days before the start of treatment or planned live attenuated vaccine vaccination during the study period;
* Had participated in other anti-tumor drug clinical trials within 4 weeks before the first drug use, and only those who had not used drugs were not subject to the 4-week time limit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) evaluated by the Independent Review Committee (IRC) | up to 33 months
  Random to the time of disease progression or death.

SECONDARY OUTCOMES:
Progression-free survival (PFS) evaluated by researcher | up to 33 months
  Random to the time of disease progression or death.
Overall survival (OS) | About 5 years
  Time from random to death.
Objective mitigation rate (ORR) | up to 33 months
  The proportion of patients whose tumor volume shrinks to the predetermined value and can maintain the minimum time limit is the sum of the proportion of complete remission (CR) and partial remission (PR).
Remission duration (DOR) | up to 33 months
  The period when the first judgment is complete or partial remission until it is found to be the progress of the disease.
Disease control rate | up to 33 months
  The number of cases with remission (PR+CR) and disease stability (SD) after treatment as a percentage of the number of evaluable cases.
No progress survival PFS rate in 12 or 24 months | up to 33 months
  If the tumor progresses or dies in 12 or 24 months, the time is from the beginning of the follow-up to the event. The proportion of all subjects who have not yet occurred at a certain time is called (no progress) survival rate.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangxi Medical University Cancer Hospital, Nanjing, Guangxi
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University cancer hospital, Harbin, Heilongjiang
  - AnYang Tumor Hospital, Anyang, Henan
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanxi Provincial Cancer Hpspital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Second People's Hospital of Neijiang, Neijiang, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Chest Hospital, Capital Medical University, Beijing

REFERENCES:
- [Derived] Liu X, Yin X, Zhuang L, Wen J, Wei Z, Cui W, Yu M, Zhao K, Liu L, Kong L, Jiang L, Jing X, Zhu H, Wang X, Dong X, Yu J, Meng X. Efficacy and safety of TQB2450 combined with anlotinib as maintenance therapy for LS-SCLC after definitive concurrent or sequential chemoradiotherapy: a prospective phase Ib study. BMC Cancer. 2025 Mar 20;25(1):509. doi: 10.1186/s12885-025-13885-8. PMID 40114144